CLINICAL TRIAL: NCT04967911
Title: Effects of Propioceptive Neuromuscular Facilitation Technique on Shoulder Pain in Paraplegic Manual Wheel Chair Users After Spinal Cord Injury
Brief Title: Effects of PNF on Shoulder Pain in Paraplegic Manual Wheel Chair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0205 Hira
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Shoulder Impingement
Keywords: Spinal cord injury, wheelchair users, Shoulder pain, PNF
MeSH Terms: conditions — Shoulder Impingement Syndrome; Spinal Cord Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic stabilization exercises (Experimental): baseline physical therapy conventional treatment along Rhythmic stabilization exercises
  Interventions: Other: Rhythmic stabilization exercises
- Conventional treatment (Other): Baseline physical therapy conventional treatment
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Rhythmic stabilization exercises — PNF techniques and Conventional Treatment:
  Experimental group received rhythmical Stabilization Technique on shoulder joint on all shoulder movements up to 1 minute in supine position For stability of joint ,re-establish dynamic rotator cuff stability and to enhance MS strength and decrease pain.
  Conventional Treatment: heating pad for 15 minutes, TENS (Transcutaneous Electrical Nerve Stimulation) and after that shoulder stretching of upper trapezius muscle, pectorals and levator scapule and isometric exercises of rotator cuff muscles performed in supine .( 10 sec hold and 10 to 15 reps)..
  Arms: Rhythmic stabilization exercises
Other: conventional treatment — Conventional Treatment: heating pad for 15 minutes, TENS (Transcutaneous Electrical Nerve Stimulation) and after that shoulder stretching of upper trapezius muscle, pectorals and levator scapule and isometric exercises of rotator cuff muscles performed in supine .( 10 sec hold and 10 to 15 reps)..
  Arms: Conventional treatment

SUMMARY:
This project was a Randomized control trial conducted to check the Effects of Proprioceptive Neuromuscular Facilitation on Shoulder Pain due to chronic impingement syndrome in paraplegic Manual Wheelchair users after Spinal Cord Injury so that we can have best treatment option for patients with shoulder pain due to manual wheelchair usage. duration was of 6months,convenient sampling was done, subject following eligibility criteria from Spine welfare trust center, Nawaz Sharif social security Hospital were randomly allocated in two groups via lottery method, Group A participants were given baseline treatment along with PNF exercises , Group B participants were given baseline treatment upto 6 weeks and 3 sessions per, post intervention assessment was done after 6 weeks, by self-generated questionnaire (WUSPI) wheel chair users shoulder pain index, (SRQ) Shoulder rating questionnaire and physical assessment by 2 special test was done, data was analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
In paraplegic manual wheelchair users Shoulder pain is most common problem after spinal cord injury. Due to wheelchair propulsion, weight relief task and other household activities repetitive load induced on upper limb and put substantial load in particular on shoulder.In spinal cord injured patients shoulder pain is because of over use of upper limb and shoulder during wheelchair related activities and personal care activities. less stability and slight muscle mass leads toward pain in their life at some point because of Muscular imbalance and later on shoulder secondary impingement syndrome. This study compared the rhythmic stabilization technique from PNF exercises with conventional treatment on experimental and control group to see the difference in reduction of pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old paraplegic manual wheel chair users after spinal cord injury.
* Those having level of injury from C7-T12
* Patients who are using wheelchair from more than one year.
* Pain perceived region of one or both Shoulder from last three months or more
* Pain without radicular symptoms radiating to whole upper limbs.
* Wheelchair propulsion in activities of daily living,
* Individuals with positive Neer's test and Hawkins-Kennedy test

Exclusion Criteria:

* Any red flags (tumor, fracture, metabolic diseases, rheumatoid arthritis, resting blood pressure greater than 140/90 mmHg, prolonged history of steroid use, etc.
* Any dislocation ,muscular tear and acute problem of shoulder.
* Presented with a diagnosis of cervical spinal stenosis, exhibited bilateral upper extremity symptoms
* Any recent surgery of the shoulder
* Individuals using other mobility devices with wheelchair.
* Individuals with primary impingement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Wheelchair User's Shoulder Pain Index | 6th Week
  The Wheelchair User's Shoulder Pain Index (WUSPI) was designed to measure shoulder pain in individuals who use wheelchairs. On the visual analog scale from ' 0' to '10 ' estimate level of pain with different activities

SECONDARY OUTCOMES:
Shoulder rating Questionnaire | 6th Week
  Shoulder rating questionnaire (SRQ) was designed to assess the severity of symptoms related to and the functional status of the shoulder. It includes domains of global assessment, pain, daily activities, recreational and athletic activities, work, satisfaction, and areas for improvement. Each domain is graded separately and is weighted to arrive at the total score

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Ikram, MS, Principal Investigator — Riphah International University
Locations (1):
- Mansoora hospital, Lahore, Spine welfare centre, Social security hosital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mason B, Warner M, Briley S, Goosey-Tolfrey V, Vegter R. Managing shoulder pain in manual wheelchair users: a scoping review of conservative treatment interventions. Clin Rehabil. 2020 Jun;34(6):741-753. doi: 10.1177/0269215520917437. Epub 2020 May 12. PMID 32397819
- [Background] El Essi K, El-Shafie JM, Al Hawamdah Z, Zaqout SI. Shoulder Pain among Rehabilitated Spinal Cord Injured Persons Using Manually Propelled Wheelchairs in the Gaza Strip: A Survey. Disabil CBR Incl Dev. 2012;23(2):53-71.
- [Background] Soo Hoo J. Shoulder Pain and the Weight-bearing Shoulder in the Wheelchair Athlete. Sports Med Arthrosc Rev. 2019 Jun;27(2):42-47. doi: 10.1097/JSA.0000000000000241. PMID 31046007
- [Background] Jain NB, Higgins LD, Katz JN, Garshick E. Association of shoulder pain with the use of mobility devices in persons with chronic spinal cord injury. PM R. 2010 Oct;2(10):896-900. doi: 10.1016/j.pmrj.2010.05.004. PMID 20970758
- [Background] Samuelsson KA, Tropp H, Gerdle B. Shoulder pain and its consequences in paraplegic spinal cord-injured, wheelchair users. Spinal Cord. 2004 Jan;42(1):41-6. doi: 10.1038/sj.sc.3101490. PMID 14713943
- [Background] Walford SL, Requejo PS, Mulroy SJ, Neptune RR. Predictors of shoulder pain in manual wheelchair users. Clin Biomech (Bristol). 2019 May;65:1-12. doi: 10.1016/j.clinbiomech.2019.03.003. Epub 2019 Mar 6. PMID 30927682
- [Background] Giner-Pascual M, Alcanyis-Alberola M, Millan Gonzalez L, Aguilar-Rodriguez M, Querol F. Shoulder pain in cases of spinal injury: influence of the position of the wheelchair seat. Int J Rehabil Res. 2011 Dec;34(4):282-9. doi: 10.1097/MRR.0b013e32834a8fd9. PMID 21971486
- [Background] Çitaker S, Taşkiran H, Akdur H, Arabaci ÜmÖ, Ekici G. Comparison of the mobilization and proprioceptive neuromuscular facilitation methods in the treatment of shoulder impingement syndrome. Pain Clin. 2005 Jun;17(2):197-202.
- [Background] Mulroy SJ, Thompson L, Kemp B, Hatchett PP, Newsam CJ, Lupold DG, Haubert LL, Eberly V, Ge TT, Azen SP, Winstein CJ, Gordon J; Physical Therapy Clinical Research Network (PTClinResNet). Strengthening and optimal movements for painful shoulders (STOMPS) in chronic spinal cord injury: a randomized controlled trial. Phys Ther. 2011 Mar;91(3):305-24. doi: 10.2522/ptj.20100182. Epub 2011 Feb 3. PMID 21292803